CLINICAL TRIAL: NCT01685333
Title: Phase 1 Assessment of Pharmacokinetics and Pharmacodynamics of Two Epoetin Alfa, Human Recombinant Epoetin (Blau Farmacêutica) and Eprex (Janssen-Cilag), After Single Dose, Intravenous Administration in Healthy Subjects: a Randomized Crossover Study.
Brief Title: PK and PD Crossover Study After Single Dose, Intravenous Administration of Two Epoetin Alfa, Human Recombinant Epoetin and Eprex, in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EPOBLA0512IV-I2; Version 1 31/05/2012 (Other: LAL Clinica)
Record Dates: First submitted 2012-07-25; First posted 2012-09-14 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Healthy
Keywords: subject
MeSH Terms: interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Other): First Period: Test Drug (Epoetin Alfa) Second Period: Comparator Drug
  Interventions: Drug: Epoetin Alfa
- Group B (Other): First period: Comparator drug Second Period: Test drug (Epoetin alfa)
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin Alfa — Intravenous single-dose administration of 100 IU/kg of the test drug (Human Recombinant Epoetin) in the first period and intravenous single-dose administration of 100 IU/kg of the comparator drug (Eprex) in the second period, after 23-30 days of washout, or vice-versa.
  Other Names: Eprex

SUMMARY:
The hypothesis of this trial is that the test drug (Eritromax ®) pharmacokinetics and pharmacodynamics parameters are similar to the comparator drug (Eprex ®) in healthy subjects following administration of single intravenous dose. The objective of this randomized, crossover, clinical trial is to evaluate the pharmacokinetic and pharmacodynamic profile of the drug Eritromax® marketed by Blau Farmacêutica, compared to the product Eprex ®, produced by Janssen-Cilag, by assessing plasma concentration of the drug and the reticulocyte count following a single-dose intravenous administration of 100 IU/kg in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Agree to all the purposes of the study by signing and dating the Informed Consent;
* Male, aged between 20 and 55 years, clinically healthy;
* BMI between 18.5 and 30;
* Hemoglobin between 13.8 and 15.4 g / dL and hematocrit between 41% and 49%;
* VCM between 82 and 98, HBMC between 26 and 34, platelets between 150,000 and 400,000 units per mL. and WBC between 3,500 to 10,500 units per ml and no atypical cells.
* Human serum ferritin between 36-262 mcg / L;
* Counting of reticulocytes in peripheral blood ≤ 3%;
* Serum erythropoietin < 30 mIU / mL.

Exclusion Criteria:

* Participation in clinical trials in the 12 months preceding the survey;
* Body weight > 100 kg;
* Presence of iron deficiency anemia;
* Presence of pulmonary, cardiovascular, neurological, endocrine, gastrointestinal, genitourinary or other systems diseases;
* Acute disease in the period of 07 days before the beginning of the practical phase (administration of the drug) of the study;
* Chronic administration of medications for hypertension, diabetes or any other disease that requires continuous use of any drug;
* Hormone therapy in the period of 02 months preceding the beginning of the practical phase (administration of the drug) of the study;
* Administration of any drug in the 02 weeks prior to the start of the practical period of the study;
* Clinical history of autoimmune or hereditary anemia;
* Clinical history of chronic bleeding;
* Clinical history of acute bleeding in the 30 days preceding the beginning of practical phase of the study (administration of the drug);
* Clinical history of allergy of biological products derived from mammalian albumin or any component of the formulation;
* Current or previous history (less than 12 months) of illicit drug abuse and / or tobacco and / or alcohol or having consumed alcohol within 48 hours prior to the practical study periods (administration of the drug);
* Prior therapies with erythropoietin;
* Albumin below 3.5 g/dL or higher than 4.8 g/dL;
* Signs or clinical history of bone marrow aplasia;
* History and clinical or laboratory liver disease;
* History and clinical or laboratory nephropathy;
* Principal Investigator of the study criteria.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-02-28 (Actual); Primary Completion 2013-10-31 (Actual); Study Completion 2013-10-31 (Actual)

PRIMARY OUTCOMES:
rHuEPO serum concentration | 1, 8, 15, 19, 22 and 26 days after first administration
  Time frame on days 1, 8, 19 and 22: -10min, 0h, 5min, 15min, 30min, 45min, 1,5h, 2h, 3h, 4h, 5h, 6h, 8h, 10h and 12h after administration;
  Time frame on day 26: -10min, 0h, 5min, 15min, 30min, 45min, 1,5h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h and 36h after last drug administration.
Plasma reticulocyte count | 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26 and 29 days after first administration of the drug.
  Time frame on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24 and 26: 10 minutes before drug administration.
  Time frame on day 29: 72 hours +/- 2 hours after last drug administration.

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clinica, Valinhos, São Paulo, Brazil